CLINICAL TRIAL: NCT02835313
Title: Promoting Recovery Optimization With WALKing Exercise After Stroke
Acronym: PROWALKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: University of Pennsylvania (Other); Christiana Care Health Services (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NIH 1R01HD086362-01A1
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FAST+SAM (Experimental): Subjects participate in fast walking training in combination with a step activity monitoring program
  Interventions: Behavioral: FAST+SAM
- FAST alone (Active Comparator): Subjects participate in fast walking training
  Interventions: Behavioral: FAST alone
- SAM alone (Active Comparator): Subjects participate in a step activity monitoring program
  Interventions: Behavioral: SAM alone

INTERVENTIONS:
Behavioral: FAST alone — Subjects participate in fast walking training 3x/week for 12 weeks.
  Arms: FAST alone
Behavioral: FAST+SAM — Subjects participate in fast walking training plus a step activity monitoring program 3x/week for 12 weeks
  Arms: FAST+SAM
Behavioral: SAM alone — Subjects participate in a step activity monitoring program 3x/week for 12 weeks
  Arms: SAM alone

SUMMARY:
Stroke survivors, as a group, are extremely inactive and this has serious consequences for them, including an increased risk of a second stroke and developing other diseases. This study investigates a novel intervention designed to improve everyday activity after stroke by combining walking training to improve walking capacity with a program to encourage more daily walking.

DETAILED DESCRIPTION:
As a group, stroke survivors are more physically inactive than even the most sedentary older adults. Lack of physical activity has serious consequences in persons with stroke, including an increased risk of recurrent stroke, developing other diseases and mortality. Current rehabilitation interventions do little to improve real-world walking activity after stroke, suggesting that simply improving walking capacity is not sufficient for improving daily physical activity after stroke. Rather, the investigator's hypothesize that the combination of a fast walking intervention that improves walking capacity, with a step activity monitoring program that facilitates translation of gains from the clinic to the "real-world", would generate greater improvements in real world walking activity than with either intervention alone. Data from the investigator's lab provides support for this hypothesis; however, it suggests that the greater efficacy of combining the 2 interventions depends on a participant's initial walking activity. Thus, the investigator's do not expect that one intervention will be superior to the others for all participants, but rather that the combined intervention will be superior for those with low levels of baseline walking activity, speed and endurance. The specific objective of this study is to test whether and for whom combining fast walking training with a step activity monitoring program (FAST+SAM) is superior in improving real-world walking activity compared to fast walking training alone (FAST) or a step activity monitoring and feedback program alone (SAM) in those with chronic stroke. Using a randomized controlled experimental design, 225 chronic (> 6 months) stroke survivors, will complete 12 weeks of fast walking training (FAST), a step activity monitoring program (SAM) or a fast walking training + step activity monitoring program (FAST+SAM). Moderation of specific intervention outcomes by baseline characteristics will be evaluated to determine for whom the interventions are effective.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-85
2. Chronic stroke (>6 months post stroke)
3. Able to walk at self-selected speed without assistance from another person (assistive devices are allowed)
4. Self-selected walking speed >0.3 m/s and <1.0 m/s
5. Average steps/day <8,000
6. Resting heart rate between 40-100 beats per minute
7. Resting blood pressure between 90/60 to 170/90.

Exclusion Criteria:

1. Evidence of cerebellar stroke
2. Other potentially disabling neurologic conditions in addition to stroke
3. Lower limb Botulinum toxin injection <4 months earlier
4. Current participation in physical therapy
5. Inability to walk outside the home prior to the stroke
6. Coronary artery bypass graft, stent placement or myocardial infarction within past 3 months
7. Musculoskeletal pain that limits activity
8. Inability to communicate with investigators
9. score >1 on question 1b and >0 on question 1c on the NIH Stroke Scale.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-07-18; Primary Completion 2023-01 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Reisman, PT, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be deposited in the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH) repository.

REFERENCES:
- [Derived] Thompson ED, McCartney KM, Pohlig RT, Hornby TG, Kasner SE, Raser-Schramm J, Henderson CE, Wright H, Wright T, Reisman DS. Maintenance of Improvements in Walking Activity in Individuals with Chronic Stroke: Follow-Up From the PROWALKS Randomized Controlled Trial. Neurorehabil Neural Repair. 2025 Oct;39(10):779-788. doi: 10.1177/15459683251352493. Epub 2025 Jul 10. PMID 40637166
- [Derived] McCartney KM, Pohlig RT, Miller A, Thompson ED, Reisman D. Matching Clinical Profiles with Interventions to Optimize Daily Stepping in People with Stroke. medRxiv [Preprint]. 2024 Nov 15:2024.11.14.24317334. doi: 10.1101/2024.11.14.24317334. PMID 39606374
- [Derived] Thompson ED, Pohlig RT, McCartney KM, Hornby TG, Kasner SE, Raser-Schramm J, Miller AE, Henderson CE, Wright H, Wright T, Reisman DS. Increasing Activity After Stroke: A Randomized Controlled Trial of High-Intensity Walking and Step Activity Intervention. Stroke. 2024 Jan;55(1):5-13. doi: 10.1161/STROKEAHA.123.044596. Epub 2023 Dec 22. PMID 38134254
- [Derived] Thompson ED, Pohlig RT, McCartney KM, Hornby TG, Kasner SE, Raser-Schramm J, Miller AE, Henderson CE, Wright H, Wright T, Reisman DS. Increasing activity after stroke: a randomized controlled trial of highintensity walking and step activity intervention. medRxiv [Preprint]. 2023 Aug 9:2023.03.11.23287111. doi: 10.1101/2023.03.11.23287111. PMID 37609269
- [Derived] Andreasen SC, Wright TR, Crenshaw JR, Reisman DS, Knarr BA. Relationships of Linear and Non-linear Measurements of Post-stroke Walking Activity and Their Relationship to Weather. Front Sports Act Living. 2020 Nov 3;2:551542. doi: 10.3389/fspor.2020.551542. eCollection 2020. PMID 33345115
- [Derived] Wright H, Wright T, Pohlig RT, Kasner SE, Raser-Schramm J, Reisman D. Protocol for promoting recovery optimization of walking activity in stroke (PROWALKS): a randomized controlled trial. BMC Neurol. 2018 Apr 12;18(1):39. doi: 10.1186/s12883-018-1044-1. PMID 29649992

RESULTS

PARTICIPANT FLOW:
Groups:
- FAST Alone: Subjects participate in fast walking training
  FAST: Subjects participate in fast walking training 3x/week for 12 weeks.
- SAM Alone: Subjects participate in a step activity monitoring program
  SAM: Subjects participate in a step activity monitoring program 3x/week for 12 weeks.
Period: Overall Study
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Started | 80 | 89 | 81
Completed POST (3-month) | 63 | 69 | 68
Completed 6-month | 62 | 68 | 58
Completed 12-month | 48 | 64 | 49
Completed | 48 | 64 | 49
Not Completed | 32 | 25 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FAST+SAM | FAST Alone | SAM Alone | Total
Number analyzed (Participants) | 80 | 89 | 81 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13.07) | 63 (11.96) | 62 (12.91) | 63 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 39 | 116
  Male | 44 | 48 | 42 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 2 | 10
  Not Hispanic or Latino | 77 | 84 | 79 | 240
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — In the study, participants self-identified their race in non-exclusive categories (e.g., they were permitted to choose "more than one race" as well as other categories). This is the format in which the data are published. Due to the constraints of this database, race data have been converted to mutually exclusive categories (e.g., an individual identifying as "more than one race" was not classified here as being in any other race category, even if the participant themselves chose other race categories.)
  Participants
    American Indian or Alaskan Native | 0 | 1 | 0 | 1
    Asian | 4 | 7 | 2 | 13
    Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 20 | 20 | 26 | 66
    White | 49 | 55 | 48 | 152
    More than one race | 6 | 5 | 5 | 16
    Unknown or not reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 80 | 89 | 81 | 250
Time since stroke [Mean (Standard Deviation); unit: months] | 42 (48.75) | 46 (62.25) | 46 (73.22) | 45 (62.04)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.13 (5.45) | 29.79 (6.39) | 31.58 (7.05) | 30.48 (6.35)
Side of hemiparesis [Count of Participants; unit: Participants]
  Left | 39 | 43 | 42 | 124
  Right | 37 | 43 | 34 | 114
  Both affected | 4 | 3 | 5 | 12
Ambulatory assistive device use [Count of Participants; unit: Participants] | 36 | 46 | 47 | 129
Lower extremity orthotic use [Count of Participants; unit: Participants] | 22 | 21 | 25 | 68
Steps per day [Mean (Standard Deviation); unit: steps/day] | 3768 (2074) | 3959 (2021) | 3845 (2193) | 3861 (2088)
Six-minute walk test distance [Mean (Standard Deviation); unit: meters] | 283 (122) | 296 (113) | 279 (110) | 287 (115)
Self-selected gait speed [Mean (Standard Deviation); unit: meters/sec] | 0.68 (0.22) | 0.71 (0.20) | 0.68 (0.22) | 0.69 (0.21)
VO2 at ventilatory threshold [Mean (Standard Deviation); unit: mL/kg per min] | 9.63 (3.35) | 8.77 (2.98) | 9.37 (2.66) | 9.24 (3.02)

OUTCOME MEASURES:

1. Primary Outcome: Steps Per Day
Description: average change in steps per day between two time points, measured over at least a 3-day period for each time point
Time Frame: Change from Baseline to 3 months (Post)
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 80 | 89 | 81
steps per day | 1307 [752 to 1861] | 406 [-63 to 876] | 1542 [1014 to 2069]

2. Primary Outcome: Steps Per Day
Description: average change in steps per day between two time points, measured over at least a 3-day period for each time point
Time Frame: Change from 3 months (Post) to 6 months
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
steps per day | -400 [-990 to 190] | -160 [-697 to 376] | -1016 [-1546 to -485]

3. Primary Outcome: Steps Per Day
Description: average change in steps per day between two time points, measured over at least a 3-day period for each time point
Time Frame: Change from 3 months (Post) to 12 months
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
steps per day | -568 [-1185 to 48] | -610 [-1162 to -59] | -1072 [-1675 to -469]

4. Secondary Outcome: Six-minute Walk Test Distance
Description: change between two time points in endurance (measured by distance attained on the 6 minute walk test)
Time Frame: Change from Baseline to 3 months (Post)
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 80 | 89 | 81
meters | 39 [23 to 56] | 43 [32 to 54] | 25 [13 to 36]

5. Secondary Outcome: Six-minute Walk Test Distance
Description: change between two time points in endurance (measured by distance attained on the 6 minute walk test)
Time Frame: Change from 3 months (Post) to 6 months
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
meters | -13 [-24 to -2] | -10 [-21 to -1] | -15 [-30 to 1]

6. Secondary Outcome: Six-minute Walk Test Distance
Description: change between two time points in endurance (measured by distance attained on the 6 minute walk test)
Time Frame: Change from 3 months (Post) to 12 months
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
meters | -18 [-32 to -3] | -21 [-33 to -9] | -16 [-32 to 1]

7. Secondary Outcome: Self-selected Gait Speed
Description: change between two time points in average self-selected speed on the 10m walk test
Time Frame: Change from Baseline to 3 months (Post)
Measure: Mean (95% Confidence Interval); unit: meters/sec
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 80 | 89 | 81
meters/sec | 0.14 [0.10 to 0.17] | 0.13 [0.10 to 0.17] | 0.11 [0.08 to 0.14]

8. Secondary Outcome: Self-selected Gait Speed
Description: change between two time points in average self-selected speed on the 10m walk test
Time Frame: Change from 3 months (Post) to 6 months
Measure: Mean (95% Confidence Interval); unit: meters/sec
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
meters/sec | -0.02 [-0.05 to 0.01] | -0.03 [-0.06 to 0.01] | -0.02 [-0.05 to 0.01]

9. Secondary Outcome: Self-selected Gait Speed
Description: change between two time points in average self-selected speed on the 10m walk test
Time Frame: Change from 3 months (Post) to 12 months
Measure: Mean (95% Confidence Interval); unit: meters/sec
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
meters/sec | -0.02 [-0.05 to 0.02] | -0.05 [-0.07 to -0.02] | -0.04 [-0.08 to 0.01]

10. Secondary Outcome: Oxygen Consumption
Description: change between two time points in average oxygen consumption at ventilatory threshold
Time Frame: Change from Baseline to 3 months (Post)
Measure: Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 80 | 89 | 81
mL/kg/min | 0.31 [-0.52 to 1.13] | 0.27 [-1.05 to 0.50] | 0.01 [-0.73 to 0.71]

11. Secondary Outcome: Oxygen Consumption
Description: change between two time points in average oxygen consumption at ventilatory threshold
Time Frame: Change from 3 months (Post) to 6 months
Measure: Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
mL/kg/min | -0.32 [-1.00 to 0.36] | -0.53 [-1.28 to 0.23] | 0.13 [-0.38 to 0.65]

12. Secondary Outcome: Oxygen Consumption
Description: change between two time points in average oxygen consumption at ventilatory threshold
Time Frame: Change from 3 months (Post) to 12 months
Measure: Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
Number analyzed (Participants) | 63 | 69 | 68
mL/kg/min | -0.08 [-1.01 to 0.86] | -1.32 [-2.06 to -0.59] | -0.15 [-0.95 to 0.66]

ADVERSE EVENTS:
Time Frame: Events separated into those occurring from randomization through post-intervention (Post - approximately 3 months) and from post-intervention (Post) up to 12 months.
Description: Systematic - regularly assessed at study appointments and scheduled phone follow-ups.
Arm/Group | FAST+SAM | FAST Alone | SAM Alone
All-Cause Mortality (participants affected / at risk) | 0/80 | 1/89 | 0/81
Serious Adverse Events (participants affected / at risk) | 14/80 | 9/89 | 3/81
Other Adverse Events (participants affected / at risk) | 25/80 | 38/89 | 19/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAST+SAM (N=80) | FAST Alone (N=89) | SAM Alone (N=81)
Recurrent Stroke (Randomization-Post) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Randomization-Post) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
Fracture (Randomization-Post) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (Randomization-Post) (General disorders) | 6 (6) | 3 (3) | 1 (1)
Death (Randomization-Post) (General disorders) | 0 (0) | 0 (0) | 0 (0)
Significant incapacity to perform ADLs for >48 hrs (Randomization-Post) (General disorders) | 0 (0) | 0 (0) | 0 (0)
Other (General disorders) | 0 (0) | 0 (0) | 0 (0)
Recurrent Stroke (Post-12 months) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Post-12 months) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
Fracture (Post-12 months) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hospitalization (Post-12 months) (General disorders) | 6 (6) | 4 (5) | 0 (0)
Death (Post-12 months) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Significant incapacity to perform ADLs for >48 hrs (Post-12 months) (General disorders) | 0 (0) | 0 (0) | 0 (0)
Other (Post-12 months) (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAST+SAM (N=80) | FAST Alone (N=89) | SAM Alone (N=81)
Falls (Randomization-Post) (General disorders) | 8 (9) | 14 (26) | 6 (9)
Dyspnea (Randomization-Post) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Open sore/blister/cut (Randomization-Post) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Muscle pain/soreness lasting >48 hrs (Randomization-Post) (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (9) | 2 (2)
Dizziness/fainting (Randomization-Post) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diaphoresis (Randomization-Post) (General disorders) | 0 (0) | 0 (0) | 0 (0)
COVID-19 illness (Randomization-Post) (General disorders) | 2 (2) | 1 (1) | 0 (0)
Other (Randomization-Post) (General disorders) | 1 (1) | 3 (3) | 3 (3)
Falls (Post-12 months) (General disorders) | 6 (6) | 4 (6) | 4 (4)
Dyspnea (Post-12 months) (General disorders) | 0 (0) | 0 (0) | 0 (0)
Open sore/blister/cut (Post-12 months) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle pain/soreness lasting >48 hrs (Post-12 months) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Dizziness/fainting (Post-12 months) (General disorders) | 0 (0) | 2 (2) | 0 (0)
Diaphoresis (Post-12 months) (General disorders) | 0 (0) | 0 (0) | 0 (0)
COVID-19 illness (Post-12 months) (General disorders) | 0 (0) | 0 (0) | 0 (0)
Other (Post-12 months) (General disorders) | 3 (4) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT02835313/Prot_SAP_000.pdf